CLINICAL TRIAL: NCT03763669
Title: Myoinositol Supplementation, Insulin Resistance and Fetal Sonographic Parameters in Gestational Diabetes, Diet Treated: a Prospective, Randomized, Placebo-controlled Study
Brief Title: Myoinositol Supplementation, Insulin Resistance and Fetal Sonographic Parameters in Gestational Diabetes Diet Treated
Acronym: MYOGDM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Messina (Other)
Responsible Party: Principal Investigator, Francesco CORRADO, Associate Professor, University of Messina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UMessina
Record Dates: First submitted 2018-11-19; First posted 2018-12-04 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Gestational Diabetes
Keywords: Insulin resistance; Fetal sonographic parameter; Myoinositol
MeSH Terms: conditions — Diabetes, Gestational; Insulin Resistance | interventions — Inositol; Folic Acid

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to receive (n. 40) diet and folic acid (400 mcg per day) alone, or (n. 40) diet, folic acid (400 mcg per day) and myoinositol (2 g. twice a day + 50 mg alfa-lactalbumin) supplementation. The insulin sensitivity index (HOMA-IR) and fetal sonographic profile will be monitor for each patient at GDM diagnosis and after 4 and 8 weeks of treatment.
Who Masked: Participant, Care Provider
Masking Description: Placebo administered
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Pregnant women randomly assigned to receive (n. 40) diet and folic acid (400 mcg per day) and myo-inositol supplementation
  Interventions: Dietary Supplement: Myoinositol
- Control (Placebo Comparator): Pregnant women randomly assigned to receive (n. 40) only diet and folic acid (400 mcg per day)
  Interventions: Dietary Supplement: Placebo (for myoinositol)

INTERVENTIONS:
Dietary Supplement: Myoinositol — myo-inositol (2 g. twice a day)
  Other Names: Folic acid
  Arms: Intervention
Dietary Supplement: Placebo (for myoinositol) — (twice a day)
  Other Names: Folic acid
  Arms: Control

SUMMARY:
The aim of this study is to verify the beneficial effects on insulin resistance and fetal sonographic parameters of a diet supplementation of myoinositol taken during the third trimester by pregnant women affected by gestational diabetes. Participants should be randomly allocated to take either myoinositol or placebo twice/day for 8 weeks. The effect of myoinositol will be checked in blood samples (insulinemia and Homeostasis Model Assessment - Insulin Resistance "HOMA-IR") and in fetal sonographic parameters after 4 and 8 weeks from the beginning of the nutritional supplementation.

DETAILED DESCRIPTION:
Background and Aim:

Gestational diabetes mellitus (GDM) is a carbohydrate intolerance diagnosed during pregnancy that is not clearly an overt diabetes. It is characterized by an increase of the physiological insulin resistance of the pregnancy status. Myo-Inositol is an insulin sensitizing agent that ameliorate the insulin resistance. The investigators have already demonstrated that myoinositol, administered in first half of pregnancy, may reduce insulin resistance and GDM incidence in pregnant women at risk for family history, obesity and overweight . But the experiences in women affected by GDM are few and controversial. So the aim of this study is to test the effectiveness of myoinositol to ameliorate the insulin resistance in GDM patients, diet treated. Moreover the investigators would like to verify the impact of this nutritional supplementation on the fetal sonographic parameters.

Design:

The study is a randomized, prospective, placebo-controlled trial, including the first 80 consecutive gestational diabetes patients diagnosed, according to the Italian Guidelines, from November 2018 to December 2019, in the Department of Obstetric and Gynecology of Messina University (ITALY). After an informed consent participants will be randomly assigned to receive (n. 40) diet and folic acid (400 mcg per day) alone, or (n. 40) diet, folic acid (400 mcg per day) and myo-inositol (2 g. twice a day + 50 mg alfa-lactalbumin) supplementation. Multiple pregnancy or known or suspected fetal congenital abnormality had been previously excluded. The insulin sensitivity index (HOMA-IR) and fetal sonographic profile will be monitor for each patient at GDM diagnosis and after 4 and 8 weeks of treatment. The pregnant women who will delivery before the time treatment (8 weeks) or who need insulin will be excluded.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy affected by gestational diabetes

Exclusion Criteria:

* Multiple pregnancy and known or suspected fetal malformations

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Insulin resistance | Start point, and 8 weeks after
  Change from baseline to 8 weeks of HOMA-IR calculated as glycemia (mmol/L) x insulinemia (mUI/L) / 22.5

SECONDARY OUTCOMES:
Fetal sonographic parameters | Start point, 4 and 8 weeks after
  Change from baseline to 4 and 8 weeks of Biparietal diameter (cm), Femur length (cm), Abdominal circumference (cm) and Subcutaneus tissue thickness (cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics & Gynecology - Policlinico "G. Martino", Messina, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Santamaria A, Alibrandi A, Di Benedetto A, Pintaudi B, Corrado F, Facchinetti F, D'Anna R. Clinical and metabolic outcomes in pregnant women at risk for gestational diabetes mellitus supplemented with myo-inositol: a secondary analysis from 3 RCTs. Am J Obstet Gynecol. 2018 Sep;219(3):300.e1-300.e6. doi: 10.1016/j.ajog.2018.05.018. Epub 2018 May 30. PMID 29859136
- [Background] Corrado F, D'Anna R, Di Vieste G, Giordano D, Pintaudi B, Santamaria A, Di Benedetto A. The effect of myoinositol supplementation on insulin resistance in patients with gestational diabetes. Diabet Med. 2011 Aug;28(8):972-5. doi: 10.1111/j.1464-5491.2011.03284.x. PMID 21414183
- [Derived] D'Anna R, Corrado F, Loddo S, Gullo G, Giunta L, Di Benedetto A. Myoinositol plus alpha-lactalbumin supplementation, insulin resistance and birth outcomes in women with gestational diabetes mellitus: a randomized, controlled study. Sci Rep. 2021 Apr 23;11(1):8866. doi: 10.1038/s41598-021-88329-x. PMID 33893377